CLINICAL TRIAL: NCT04472585
Title: Sub-cutaneous Ivermectin in Combination With and Without Oral Zinc: a Placebo Randomized Control Trial on Mild to Moderate COVID-19 Patients
Brief Title: Efficacy of Subcutaneous Ivermectin With or Without Zinc in COVID-19 Patients
Acronym: SIZI-COVID-PK
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sohaib Ashraf (Other)
Responsible Party: Sponsor-Investigator, Sohaib Ashraf, Post-Graduate Resident Cardiology, Sheikh Zayed Federal Postgraduate Medical Institute
Organization: Sheikh Zayed Federal Postgraduate Medical Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SZMC/IRB/Internal/215/2020
Record Dates: First submitted 2020-07-14; First posted 2020-07-15 (Actual); Last update posted 2021-02-17 (Actual); Status verified 2021-02

CONDITIONS: Coronavirus Infection; COVID; Sars-CoV2
Keywords: SARS-Cov-2; COVID-19; Coronavirus; Ivermectin; Zinc
MeSH Terms: conditions — Coronavirus Infections; COVID-19 | interventions — Saline Solution; Zinc; Ivermectin

STUDY DESIGN:
Intervention Model Description: randomized, controlled, multi-armed, open-label, interventional study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Empty capsule will sub-cutaneous injection of ivermectin will be used
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- Ivermectin alone (Active Comparator): Sub-cutaneous injection ivermectin 200ug/kg body weight once every 48 hourly plus standard care
  Interventions: Drug: Ivermectin Injectable Solution; Drug: Placebo empty capsule
- Ivermectin with Zinc (Active Comparator): Sub-cutaneous injection ivermectin 200ug/kg body weight once every 48 hourly with 20mg Zinc Sulphate 8 hourly plus standard care
  Interventions: Drug: Ivermectin Injectable Solution; Drug: Zinc; Drug: Placebo empty capsule
- Placebo (Placebo Comparator): Placebo drug plus standard care
  Interventions: Other: Injectable Placebo; Drug: Placebo empty capsule
- Ivermectin (oral) alone (Active Comparator): Oral ivermectin 0.2mg/kg/day
  Interventions: Drug: Placebo empty capsule; Drug: Oral Ivermectin
- Ivermectin (oral) with Zinc (Active Comparator): Oral ivermectin 0.2mg/kg/day with 20mg Zinc Sulphate 8 hourly plus standard care
  Interventions: Drug: Zinc; Drug: Placebo empty capsule; Drug: Oral Ivermectin
- Zinc Alone (Active Comparator): 20mg Zinc Sulphate 8 hourly plus standard care
  Interventions: Drug: Zinc; Drug: Placebo empty capsule

INTERVENTIONS:
Drug: Ivermectin Injectable Solution — Subcutaneous Ivermectin 200ug/kg body weight 48 hourly
  Other Names: Montpellier
  Arms: Ivermectin alone; Ivermectin with Zinc
Other: Injectable Placebo — 0.9% normal saline
  Other Names: 0.9% normal saline
  Arms: Placebo
Drug: Zinc — Zinc Sulphate 20mg 3 times a day
  Arms: Ivermectin (oral) with Zinc; Ivermectin with Zinc; Zinc Alone
Drug: Placebo empty capsule — Placebo empty capsule
Drug: Oral Ivermectin — 0.2mg/kg/day
  Arms: Ivermectin (oral) alone; Ivermectin (oral) with Zinc

SUMMARY:
To measure the effect of Ivermectin (sub-cutaneous) with or without zinc in treating the COVID-19 patients to clear viral load of SARS-CoV-2 along with reduction in severity of symptoms and length of hospitalization of patients with COVID-19.

DETAILED DESCRIPTION:
This is a parallel assigned, randomized, controlled, multi-armed, investigator Initiated interventional study is designed to demonstrate efficacy to lower the viral load of COVID-19 and to demonstrate the antiviral effects of subcutaneous Ivermectin with or without zinc in mild to moderate symptomatic patients who consent to randomization following a new diagnosis in Pakistan with COVID-19 (PCR positive). Investigators will follow up with participants daily and PCR will be done on alternate days in BSL-3 lab. Dose will only be repeated if test remained positive..

ELIGIBILITY:
Inclusion Criteria:

* Nasopharyngeal RT-PCR positive SARS-CoV-2 patient with mild to moderate disease
* Age 18 and above
* BMI 18-28 kg/m

Exclusion Criteria:

* Allergy to any drug
* Co-morbidities: any pre-existing cardiac disease, pulmonary disease
* Arrhythmias
* Pregnancy
* RT-PCR performed >3 days prior to enrollment

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 180 (Estimated)
Dates: Start 2020-11-14 (Actual); Primary Completion 2021-08-15 (Estimated); Study Completion 2021-10-30 (Estimated)

PRIMARY OUTCOMES:
qRT-PCR | 14 days
  time needed to turn positive COVID-19 PCR to negative
Time taken for alleviation of symptoms | upto 14 days
  time needed to turn off symptoms
Severity of symptoms | upto 14 days
  time needed of symptom serverity

SECONDARY OUTCOMES:
Severity of symptoms | 14 days
  time needed to make patients clinically better
Morality | 30 days
  death rate

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Ashraf, PhD, Study Chair — University of Veterinary & Animal Sciences, Lahore, Pakistan; Shoaib Ashraf, PhD, Study Director — Harvard University Boston, USA; Sohaib Ashraf, MBBS, Principal Investigator — Shaikh Zayed Medical Complex, Pakistan; Moneeb Ashraf, MBBS, Principal Investigator — Mayo Hospital, Pakistan
Locations (2):
- Pakistan (2):
  - Ali Clinic, Lahore, MA
  - Shaikh Zayed Hospital, Lahore, Punjab Province

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Simsek Yavuz S, Unal S. Antiviral treatment of COVID-19. Turk J Med Sci. 2020 Apr 21;50(SI-1):611-619. doi: 10.3906/sag-2004-145. PMID 32293834
- [Background] Patri A, Fabbrocini G. Hydroxychloroquine and ivermectin: A synergistic combination for COVID-19 chemoprophylaxis and treatment? J Am Acad Dermatol. 2020 Jun;82(6):e221. doi: 10.1016/j.jaad.2020.04.017. Epub 2020 Apr 10. No abstract available. PMID 32283237
- [Background] Caly L, Druce JD, Catton MG, Jans DA, Wagstaff KM. The FDA-approved drug ivermectin inhibits the replication of SARS-CoV-2 in vitro. Antiviral Res. 2020 Jun;178:104787. doi: 10.1016/j.antiviral.2020.104787. Epub 2020 Apr 3. PMID 32251768
- [Derived] Ashraf S, Ashraf S, Farooq I, Ashraf S, Ashraf M, Imran MA, Kalsoom L, Akmal R, Ghufran M, Rafique S, Akram MK, Habib Z, Siddiqui UN, Ahmad A, Arshad S, Virk MAR, Gul M, Awais AB, Hassan M, Sherazi SSH, Safdar Z, Munir I, Khalid H, Munir K, Majeed N, Alahmadi YM, Humayun A, Saboor QA, Ahmad A, Ashraf M, Izhar M; DOCTORS LOUNGE Consortium. Anti-COVID property of subcutaneous ivermectin in synergy with zinc among midlife moderately symptomatic patients: a structured summary of a study protocol for a randomised controlled trial. Trials. 2021 Sep 6;22(1):591. doi: 10.1186/s13063-021-05487-z. PMID 34488858